CLINICAL TRIAL: NCT06931964
Title: The Level of Frailty in Individuals Diagnosed With Primary Sarcopenia; Balance, Fall Risk and Impact on Kinesiophobia
Brief Title: Frailty and Assocciated Factors in Sarcopenia
Status: Completed | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, METEHAN YANA, Supervisor, PhD, Karabuk University
Other Study IDs: Karabuk 001
Record Dates: First submitted 2025-02-11; First posted 2025-04-17 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sarcopenia: According to EWGSOP2 criteria; individuals diagnosed with sarcopenia were included in the study by evaluating low muscle strength, low muscle quantity or quality, and low physical performance.

SUMMARY:
Primary sarcopenia is a condition that occurs with the aging process and is characterized by symptoms such as decreased muscle mass, impaired muscle function and decreased physical strength. The decrease in muscle mass can lead to a decrease in physical strength, balance and mobility, making older people more prone to frailty and falls, which can lead to a fear of falling. Although there are few studies on sarcopenia in the literature, the level of frailty in sarcopenia is related to balance, falls risk and kinesiophobia in sarcopenia.

Our aim in the study was to measure frailty in elderly individuals diagnosed with sarcopenia and to determine the level of frailty.

to evaluate the effect of sarcopenia on fall risk, balance and kinesiophobia and to evaluate the effect of sarcopenia on fall risk, balance and kinesiophobia according to the results of the evaluation and new rehabilitation programs on frailty, falls, kinesiophobia and balance resulting from sarcopenia and to be the basic data for the programs to be created.

DETAILED DESCRIPTION:
Primary sarcopenia is a condition that occurs with the aging process and is characterized by symptoms such as decreased muscle mass, impaired muscle function and decreased physical strength. The decrease in muscle mass can lead to a decrease in physical strength, balance and mobility, making older people more prone to frailty and falls, which can lead to a fear of falling. Recent studies have shown that sarcopenia is closely related to frailty. Frailty is a clinical syndrome characterized by decreased strength, endurance and physiological function, including dysregulation of immune, endocrine, stress and energy regulation systems, which can make individuals more prone to physical dysfunction, loss of balance and falls. Sarcopenia can cause balance problems as it leads to muscle weakness and loss. Lack of balance puts individuals at risk of falling while performing activities of daily living increases. The risk of falling is a major concern for individuals with sarcopenia. Factors such as muscle weakness, poor balance and coordination increase the risk of falls. Kinesiophobia is frequently observed in individuals with sarcopenia. Kinesiophobia refers to the fear or avoidance of movement. Sarcopenia can limit individuals' mobility and they may develop kinesiophobia due to pain while performing daily activities or fear of falling. Kinesiophobia can limit individuals' active lifestyle and further reduce their physical functioning. As a result, the level of frailty in individuals with sarcopenia may have a negative impact on balance, fall risk and kinesiophobia. There is no study in the literature that includes the effect of frailty level on balance, fall risk and kinesiophobia in primary sarcopenia. With this study, the investigators aim to fill this gap in the literature by examining the effect of frailty level on balance, fall risk and kinesiophobia. As a common effect, the investigators think that the results of our study can be used in rehabilitation programs aiming to improve functional levels in individuals diagnosed with primary sarcopenia. It will contribute to the correct evaluation of activity and participation limitations, determination of priorities, selection of the right activity in treatment approaches, and more effective results when adapted with technology-supported approaches.

ELIGIBILITY:
Inclusion criteria:

1. Volunteering to participate in the study
2. 65 years of age or older
3. Being diagnosed with primary sarcopenia by a specialist
4. To have the cooperation to perform the measurements

Exclusion criteria:

1. Having a disease that will affect balance (vertigo etc.)
2. Not volunteering to participate in the study
3. History of trauma within the last six months (fracture, soft tissue injury, etc.)
4. Having undergone lower extremity surgery

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients with sarcopenia included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Frailty | Baseline
  Frailty will be assessed with the Edmonton Frailty Scale. It is scored between 0-17. Frailty increases as the score increases. 0-4 points: Not frail, 5-6 points: Mildly frail, 7-8 points: Moderately frail, 9-17 points: Severely frail.
Risk of falling | Baseline
  Fall risk will be assessed with the Denn Fall Risk Assessment Scale. The total score is generally: 0-3: Low risk, 4-6: Medium risk, 7 and above: High risk.
Kinesiophobia | Baseline
  The Tampa Kinesiophobia Scale will be used to assess kinesiophobia. Total score: 17-68. Higher scores indicate greater kinesiophobia (fear of movement).
Balance | Baseline
  Balance will be assessed with a posturography device.

CONTACTS AND LOCATIONS:
Overall Officials: Metehan Yana, Principal Investigator — Karabuk University; Ecem Çoroğlu, BD, Principal Investigator — Karabuk University
Locations (1):
- Karabük University, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ye L, Liang R, Liu X, Li J, Yue J, Zhang X. Frailty and sarcopenia: A bibliometric analysis of their association and potential targets for intervention. Ageing Res Rev. 2023 Dec;92:102111. doi: 10.1016/j.arr.2023.102111. Epub 2023 Oct 29. PMID 38031836
- [Result] Alvarez-Bustos A, Carnicero-Carreno JA, Davies B, Garcia-Garcia FJ, Rodriguez-Artalejo F, Rodriguez-Manas L, Alonso-Bouzon C. Role of sarcopenia in the frailty transitions in older adults: a population-based cohort study. J Cachexia Sarcopenia Muscle. 2022 Oct;13(5):2352-2360. doi: 10.1002/jcsm.13055. Epub 2022 Jul 28. PMID 35903871